CLINICAL TRIAL: NCT02460640
Title: The Effects of Ultrasound-guided Transversus Abdominis Plane Block on Acute and Chronic Postsurgical Pain After Robotic Partial Nephrectomy. A Prospective, Randomized, Clinical Trial
Brief Title: The Effects of TAP Block on Postsurgical Pain After Minimally Invasive Partial Nephrectomy:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, Head of Anestesiology and Critical Care Department, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tap Block
Record Dates: First submitted 2015-05-19; First posted 2015-06-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Acute Pain; Chronic Pain
Keywords: Minimally invasive surgery; Partial nephrectomy
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Analgesia, Patient-Controlled; Morphine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tap Block (Active Comparator): the intervention will be tap block after induction of anesthesia with ropivacaine 0,5% 15ml and continuous patient-controlled analgesia with morphine
  Interventions: Procedure: Tap block; Procedure: intravenous Patient controlled analgesia; Drug: Morphine; Drug: Ropivacaine
- No Tap Block (Active Comparator): the patients who not receive tap block but they will be as intervention intravenous Patient controlled analgesia
  Interventions: Procedure: intravenous Patient controlled analgesia; Drug: Morphine

INTERVENTIONS:
Procedure: Tap block — intravenous patient-controlled analgesia with morphine and tap block with subcostal and posterior approach with ropivacaine 0,5% 15ml+15ml
  Arms: Tap Block
Procedure: intravenous Patient controlled analgesia — intravenous patient-controlled analgesia with morphine
Drug: Morphine
Drug: Ropivacaine
  Arms: Tap Block

SUMMARY:
Single-center study in order to assess whether the tap block can make extremely beneficial in terms of reducing the acute and chronic pain as well as for use of opioids and side effects related to it in patients undergoing surgery to minimally invasive partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* asa score I,II,II
* patients scheduled for robot assisted partial nephrectomy

Exclusion Criteria:

* previous abdominal surgery
* inability to provide informed consent
* allergy to the anesthetic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Morphine consuption 24 hr after surgery | 24 hours
  Cumulative morphine consuption (mg) 24 hr starting from the time of extubation.
Acute pain after surgery measured with Numerical Rating Scale | 24 hours
  patients were assessed for pain, according to Numerical Rating Scale (NRS; 0: no pain to 10: worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena CI, Rome, Italy

REFERENCES:
- [Derived] Covotta M, Claroni C, Costantini M, Torregiani G, Pelagalli L, Zinilli A, Forastiere E. The Effects of Ultrasound-Guided Transversus Abdominis Plane Block on Acute and Chronic Postsurgical Pain After Robotic Partial Nephrectomy: A Prospective Randomized Clinical Trial. Pain Med. 2020 Feb 1;21(2):378-386. doi: 10.1093/pm/pnz214. PMID 31504875